CLINICAL TRIAL: NCT03728413
Title: The Impact of Age on Adaptive Immunity in Adults Infected With Respiratory Syncytial Virus
Acronym: INFLAMMAGE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 14SM2070
Record Dates: First submitted 2018-10-16; First posted 2018-11-02 (Actual); Results first posted 2026-01-26 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: RSV Infection
Keywords: Elderly; Human; Respiratory Syncytial Infections; RNA Virus Infections
MeSH Terms: conditions — Respiratory Syncytial Virus Infections; RNA Virus Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Healthy, non-smoking or ex-smoking persons aged 60 to 75 years (Other): RSV A Memphis 37 will be given as intra-nasal drops.
  Interventions: Biological: RSV A Memphis 37

INTERVENTIONS:
Biological: RSV A Memphis 37 — Subjects will be inoculated using intra-nasal drops with diluted inoculum at a given dose divided equally between the two nostrils. Dose: Good Manufacturing Practices-certified RSV Memphis 37 10(4) PFU in 1ml, 25% sucrose/Dulbecco's Modification of Eagle's Medium. Inoculations using intranasal drops will be done using a 1mL pipette with subjects supine. This will be done slowly with sufficient interval between each inoculation (2-3 minutes) to ensure maximum contact time between with the nasal and pharyngeal mucosa. Subjects will be asked not to swallow during the procedure to ensure maximal pharyngeal contact.
  Following inoculation, advice regarding hand hygiene will be given, subjects will be provided with alcohol hand gel and facemasks to reduce spread of virus in the environment.

SUMMARY:
This study will for the first time systematically investigate the immune responses in an elderly cohort challenged with a well-defined RSV inoculum. With a global aging population and continuing difficulties in generating vaccines that can reliably induce protective immunity in the elderly, these data will indicate the targets at which development of vaccines against RSV and other infections should be directed.

DETAILED DESCRIPTION:
Respiratory syncytial virus (RSV) is one of the most common causes of chest infection worldwide, with 64 million episodes and 160,000 deaths each year. Despite this, it remains an underappreciated health problem and there are currently no specific treatments or vaccines against it. Although RSV infection is most frequent in young children, the majority of deaths occur in older adults, particularly in those with underlying heart and lung disease. This is believed to be due in part to the ageing immune system's reduced ability to protect against infection and symptomatic disease. However, little is known about the way human immune responses to RSV infection in older individuals differ from those of younger people. Further understanding of the mechanisms underlying immunity and potential impairments in these higher-risk people are therefore necessary. This project aims to study the role of T cells (which destroy virus-infected cells and are likely to be essential for recovery from infection) in healthy older volunteers after they have been given an RSV-induced common cold. Samples will be taken from the blood and respiratory tract in order to identify the differences in T cell responses that occur in older adults compared with their younger counterparts. Participants will be carefully screened to ensure they do not have any underlying health problems that might make them more at risk of severe disease and will be monitored closely throughout the course of infection. The investigators anticipate that T cell function even in healthy older individuals will be impaired compared to young adults, thus contributing in those with additional health problems to more severe disease. By analysing the networks of genes that are switched on and off, the investigators aim to identify the particular defects underlying these functional defects in order to ultimately define targets for novel treatments and T cell-stimulating vaccines.

ELIGIBILITY:
Inclusion Criteria:

* Healthy persons aged 60 to 75 years, able to give informed consent
* Non smokers or ex-smokers with smokers with less than or equal to 5 pack years smoking history.
* Spirometry within the normal range for age and height (+/- 15%)
* FEV1/FVC >70% pre-bronchodilator

Exclusion Criteria:

* Chronic respiratory disease (asthma, COPD, rhinitis, sinusitis) in adulthood
* Inhaled bronchodilator or steroid use within the last 12 months
* Habitual use of any medication or other product (prescription or over-the-counter) for symptoms of rhinitis or nasal congestion within the last 3 months
* Acute upper respiratory infection (URI or sinusitis) in the past 6 weeks
* Subjects with allergic symptoms present at baseline
* Clinically relevant abnormality on chest X-ray
* Those in close domestic contact (i.e. sharing a household with, caring for, or daily face to face contact) with children under 3 years, other elderly adults (>65 years), immunosuppressed persons, or those with chronic respiratory disease
* Subjects with known or suspected immune deficiency
* Receipt of systemic glucocorticoids (in a dose ≥ 5 mg prednisone daily or equivalent) within one month, or any other cytotoxic or immunosuppressive drug within 6 months prior to challenge
* Known IgA deficiency, immotile cilia syndrome, or Kartagener's syndrome
* History of frequent nose bleeds
* Any significant medical condition or prescribed drug deemed by the study doctor to make the participant unsuitable for the study
* Women of childbearing potential must have a negative hCG urine pregnancy test *
* Positive urine drug screen
* Women of childbearing potential will have a pregnancy test performed prior to virus inoculation to exclude pregnancy and be required to use contraception throughout the study.

Ages: 60 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2018-11-12 (Actual); Primary Completion 2023-05-04 (Actual); Study Completion 2023-05-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Chiu, Principal Investigator — Imperial College London
Locations (1):
- Imperial College London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
Data may be shared, all data will be anonymised.

REFERENCES:
- [Derived] Ascough S, Dayananda P, Kalyan M, Kuong SU, Gardener Z, Bergstrom E, Paterson S, Kar S, Avadhan V, Thwaites R, Sanchez Sevilla Uruchurtu A, Ruckwardt TJ, Chen M, Nair D, Derrien-Colemyn A, Graham BS, Begg M, Hessel E, Openshaw P, Chiu C. Divergent age-related humoral correlates of protection against respiratory syncytial virus infection in older and young adults: a pilot, controlled, human infection challenge model. Lancet Healthy Longev. 2022 Jun;3(6):e405-e416. doi: 10.1016/S2666-7568(22)00103-9. Epub 2022 Jun 9. PMID 36098319

RESULTS

PARTICIPANT FLOW:
Groups:
- Healthy, Non-smoking or Ex-smoking Persons Aged 60 to 75 Years: RSV A Memphis 37 will be given as intra-nasal drops to healthy, non-smoking or ex-smoking persons aged 60 to 75 years
- Healthy, Non-smoking or Ex-smoking Persons Aged 18 - 40 Years: RSV A Memphis 37 will be given as intra-nasal drops to healthy, non-smoking or ex-smoking persons aged 18 - 40 years
Period: Overall Study
Arm/Group | Healthy, Non-smoking or Ex-smoking Persons Aged 60 to 75 Years | Healthy, Non-smoking or Ex-smoking Persons Aged 18 - 40 Years
Started | 28 | 0
Completed | 28 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: We recruited 28 persons aged between 65-75years for this study. No participants between the age of 18-40 years were consented and enrolled under this protocol.
Groups:
- Healthy, Non-smoking or Ex-smoking Persons Aged 60 to 75 Years: RSV A Memphis 37 will be given as intra-nasal drops.
  RSV A Memphis 37: Subjects will be inoculated using intra-nasal drops with diluted inoculum at a given dose divided equally between the two nostrils. Dose: Good Manufacturing Practices-certified RSV Memphis 37 10(4) PFU in 1ml, 25% sucrose/Dulbecco's Modification of Eagle's Medium. Inoculations using intranasal drops will be done using a 1mL pipette with subjects supine. This will be done slowly with sufficient interval between each inoculation (2-3 minutes) to ensure maximum contact time between with the nasal and pharyngeal mucosa. Subjects will be asked not to swallow during the procedure to ensure maximal pharyngeal contact.
  Following inoculation, advice regarding hand hygiene will be given, subjects will be provided with alcohol hand gel and facemasks to reduce spread of virus in the environment.
Arm/Group | Healthy, Non-smoking or Ex-smoking Persons Aged 60 to 75 Years
Number analyzed (Participants) | 28
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 13
  >=65 years | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.46 (4.16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 20
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White British | 23
  White Irish | 1
  White Other | 2
  Black or Black British | 1
  Asian or Asian British | 1
Region of Enrollment [Number; unit: participants]
  United Kingdom | 28

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Challenge-related Adverse Events
Description: To determine the safety and tolerability of experimental challenge with RSV Memphis 37, assessed by the number of participants with challenge-related adverse events. This includes any AEs deemed at least possibly related to the study challenge intervention (RSV Memphis 37). Assessed from the time of inoculation to study completion (Day 180).
Time Frame: 180 days
Population: In the "Healthy, non-smoking or ex-smoking persons aged 60 to 75 years" arm, 28 participants were enrolled.
Measure: Count of Participants; unit: Participants
Groups:
- Healthy, Non-smoking or Ex-smoking Persons Aged 60 to 75 Years: All enrolled participants are inoculated with RSV Memphis 37. Some meet the criteria for becoming infected, while other participants resist infection i.e. are uninfected.
Arm/Group | Healthy, Non-smoking or Ex-smoking Persons Aged 60 to 75 Years
Number analyzed (Participants) | 28
Participants
  Infected: number analyzed (Participants) | 19
  Infected | 0
  Uninfected: number analyzed (Participants) | 9
  Uninfected | 3

2. Secondary Outcome: Symptom Severity in RSV Infection
Description: This is the total symptom score for the whole 14 day period and is therefore the sum of all the scores from Day 0 to Day 14.
  Self-reported upper and lower respiratory and systemic symptoms by diary card. A self-completed diary card of upper respiratory tract clinical symptoms was completed on Day 0 and daily for 14 days after inoculation.
  A total 'upper respiratory clinical symptom score' will be derived using a four-point scale (0-3 for absent, mild, moderate and severe) for each of the following four respiratory symptoms: sneezing, nasal discharge, nasal obstruction, and sore throat, giving a maximum clinical severity score of 12 per day.
Time Frame: Day 0 to Day 14 (14 days)
Population: 1 participant was excluded from analysis as they were co-infected with SARS-CoV-2 and Influenza
Measure: Median (Inter-Quartile Range); unit: Total symptom score
Arm/Group | Healthy, Non-smoking or Ex-smoking Persons Aged 60 to 75 Years
Number analyzed (Participants) | 27
Total symptom score
  Infected: number analyzed (Participants) | 18
  Infected | 2.21 [0.95 to 3.74]
  Uninfected: number analyzed (Participants) | 9
  Uninfected | 0.75 [0.38 to 0.88]

3. Secondary Outcome: Nasal Viral Load Measurement in RSV Infection
Description: Change from baseline in viral load by qPCR of 28 days post inoculation.
Time Frame: Day 0 to Day 28 (28 days)
Population: 1 participant was excluded from analysis as they were co-infected with SARS-CoV-2 and Influenza
Measure: Median (Inter-Quartile Range); unit: Nasal Viral Load (log10 copies per mL)
Arm/Group | Healthy, Non-smoking or Ex-smoking Persons Aged 60 to 75 Years
Number analyzed (Participants) | 27
Nasal Viral Load (log10 copies per mL)
  Infected: number analyzed (Participants) | 18
  Infected | 28.88 [15.62 to 44.2]
  Uninfected: number analyzed (Participants) | 9
  Uninfected | 0.00 [0.00 to 0.00]

4. Other Pre Specified Outcome: Antibody Responses to RSV Infection
Description: Mean titre of RSV specific antibodies from the Day 0, Day 7, Day 10, Day 14 and Day 28 sampling timepoints post inoculation in the infected vs uninfected group.
Time Frame: Day 0 to Day 28 (28 days)
Population: 1 participant was excluded from analysis as they were co-infected with SARS-CoV-2 and Influenza
Measure: Geometric Mean (95% Confidence Interval); unit: Anti-F protein Serum IgG titer
Arm/Group | Healthy, Non-smoking or Ex-smoking Persons Aged 60 to 75 Years
Number analyzed (Participants) | 27
Anti-F protein Serum IgG titer
  Infected: number analyzed (Participants) | 18
  Infected | 12.27 [11.29 to 13.33]
  Uninfected: number analyzed (Participants) | 9
  Uninfected | 9.55 [7.065 to 12.90]

5. Other Pre Specified Outcome: T Cell Responses to RSV Infection
Description: Frequency of RSV specific T cells measured at 0,7,10,14 and 28 days post inoculation
Time Frame: Day 0 to Day 28 (at 0,7,10,14 and 28 days post inoculation)
Population: No measurements were performed for this outcome measure.
Arm/Group | Healthy, Non-smoking or Ex-smoking Persons Aged 60 to 75 Years
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 180 days
Arm/Group | Healthy, Non-smoking or Ex-smoking Persons Aged 60 to 75 Years
All-Cause Mortality (participants affected / at risk) | 0/28
Serious Adverse Events (participants affected / at risk) | 0/28
Other Adverse Events (participants affected / at risk) | 23/28
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Healthy, Non-smoking or Ex-smoking Persons Aged 60 to 75 Years (N=28)
Hypotension (Cardiac disorders) | 4 (7)
Bleeding (Infections and infestations) | 7 (9) — Bleeding during bronchoscopy procedure
COVID-19 (Infections and infestations) | 2 (2)
Chills (Infections and infestations) | 2 (2) — Feeling of chills without pyrexia
Influenza-like-illness (Infections and infestations) | 2 (2)
Hypoxemia (Respiratory, thoracic and mediastinal disorders) | 4 (5)
Airway inflammation (Respiratory, thoracic and mediastinal disorders) | 2 (2) — Airway inflammation noted during bronchoscopy procedure
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Nausea (Gastrointestinal disorders) | 2 (3)
Pre-syncopal epiosode (Nervous system disorders) | 2 (2)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-11-01): https://cdn.clinicaltrials.gov/large-docs/13/NCT03728413/Prot_SAP_000.pdf
  • Informed Consent Form (2022-10-03): https://cdn.clinicaltrials.gov/large-docs/13/NCT03728413/ICF_001.pdf